CLINICAL TRIAL: NCT03970486
Title: Effects of Two Different Dry-Needling Techniques on Lumbar Multifidus Muscle Activation and Pressure Pain Threshold in Healthy Adults and Patients With Low Back Pain
Brief Title: Effects of Two Different Dry-Needling Techniques for Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Texas Woman's University (Other)
Collaborators: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Sharon Wang-Price, Professor, Texas Woman's University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19750
Record Dates: First submitted 2017-09-22; First posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: Participants will be assigned into two dry needling treatment groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Needle Manipulation (Active Comparator): Participant will receive dry needling intervention with manipulation.
  Interventions: Procedure: Dry needling
- In Situ (Active Comparator): Participant will receive dry needling intervention without manipulation.
  Interventions: Procedure: Dry needling

INTERVENTIONS:
Procedure: Dry needling — For the needle manipulation technique, the needle will be pulled in and out (sparrow pecking) and redirected in small angles (coning) for 5-10 seconds. For the in situ technique, the needles will stay (in situ) in the left and right lumbar multifidus muscles for 10 minutes after the insertion of the needle.

SUMMARY:
Although dry-needling with or without manipulation has shown to be a useful technique to reduce pain in patients with low back pain (LBP), it is unclear which of these two dry-needling techniques would have a greater effect on the lumboscaral multifidus (LM) muscle activation, which is essential in LBP rehabilitation. Therefore, the purposes of the study are: 1) to investigate whether or not dry-needling would change muscle activity of the LM muscles in asymptomatic healthy adults and in individuals with LBP, respectively, and 2) to compare the effects of two dry-needling techniques on LM muscle activation and pressure pain threshold (PPT) in asymptomatic healthy adults and individuals with LBP, respectively.

DETAILED DESCRIPTION:
PARTICIPANTS

Participants will be recruited from local communities, including but not limited to Texas Woman's University (TWU) via flyers. The flyers will be posted at the TWU - Dallas campus, and Texas Physical Therapy Specialist - Dallas where one of the principal investigators, Zach Couch, works, and other community centers with approval.

Participants who are interested in taking part in the study will be asked to call the investigators to schedule an appointment. The consent form will be presented at the beginning of the appointment.

Eligible participants are English-speaking adults and are 18 years of age or older. Additional criteria for asymptomatic healthy adults include no existing LBP and no LBP in the past 6 months. Additional criteria for symptomatic participants include existing LBP near the L5-S2 level with an average pain intensity score ≥ 2/10 in the past 24 hours (numeric pain rating scale of 0-10, 0 being no pain, 10 being unbearable pain).

Exclusion criteria for all participants include bleeding disorders (e.g. hemophilia), use of anti-coagulants (e.g. Coumadin), previous low back surgery, systemic joint disease (e.g. rheumatoid arthritis), cancer of the lower quadrant, neurological disorders, allergic reaction to adhesive tape, or inability to obtain the testing position (prone lying).

OUTCOME MEASURES

1. Electromyographic (EMG) activity A Delsys EMG system with 2 wireless surface electrodes (Delsys Inc., Natick, MA) will be used to obtain muscle activities of the LM, one at the L5 level, and the other at the S2 level. The bandwidth of the EMG system will be set at 20 to 450 Hz with a gain of 1,000. The EMG signal will be recorded at a sampling rate of 2,000 Hz. Each surface electrode has a built-in reference electrode.
2. Pressure Pain Threshold (PPT) A hand-held computerized pressure algometer (Medoc ltd., Ramat Yishai, Israel) will be used to determine the PPT on the two most tender points corresponding to the two EMG electrode sites. The algometer consists of a 1-cm2 round tip that will be pressed vertically on the target locations of the muscle. To provoke the patient's pain or discomfort, pressure will be increased at a rate of 40 kPa/sec until the participant feels pain as indicated by pressing a patient safety unit. The limit of pressure threshold will be set at 800 kPa, meaning that a pressure exceeding 800 kPa will be cut off to minimize tissue damage. If the participant does not push the button at 800 kPa, a value of 800 is used as the threshold value.

PROCEDURE

After participants are informed of the risks, benefits and procedures of the study, they will be asked to sign a written consent form approved by the TWU Institutional Review Board - Dallas. Eligible participants will be asked to complete an intake form to collect their demographic data (age, gender, height, weight, occupation, hand dominance), past medical history, and questions related to their past history of pain if applicable (onset, injury mechanism if any, location, duration, type, and nature). The symptomatic participants also will be asked to rate their pain intensity at present, at worst, and at best in the past 24 hours using the NPRS. Participants who exhibit any of the exclusion criteria will be excluded from the study. Once the participants is determined to be eligible for the study, they will be asked to complete the Modified Oswestry Low Back Pain Disability Questionnaire (OSW), which will be used to determine their perceived disability and functional limitations due to LBP.

Next, the EMG activity and PPTs will be collected from the painful side of the participants with LBP and the right side of the asymptomatic participants. When the symptomatic participants have bilateral LBP, the EMG activity and PPTs will be collected from the most painful side. If both sides are equally painful, a coin toss was performed to select the side (heads for the right side, tails for the left side).

During the EMG and PPT testing, participants will be asked to lie in a prone position on an examination table with their arms on the sides. A pillow was placed under the participant's abdomen to flatten the lumbar lordotic curve and an inclinometer will be placed on the lumbosacral junction to ensure the lumbar curve ≤10°. The spinous processes of the L1-S2 and posterior superior iliac spine (PSIS) will be be identified by palpation and marked with a skin marker.

1. EMG Activity Recording

   To prepare for EMG recording, each participant's skin over the LM muscles (between L4-S2) will be cleaned with alcohol and, if needed, excessive hair will be shaved using a disposable razor. Adhesive tape will be used to affix two wireless EMG electrodes to the skin over the LM muscles, one at the L5 level and the other at the S2 level. Following the recommendation by the Surface ElectroMyoGraphy for the Non-Invasive Assessment of Muscles (SENIAM) project (http://www.seniam.org/), the L5 electrodes were placed at the level of the L5 spinous process (i.e. about 2 - 3 cm from the midline) and aligned with a line from the posterior superior iliac spine (PSIS) to the interspace between the L1 and L2 spinous process. The S2 electrode was placed medial to the PSIS.

   During EMG recording, participants will be asked to abduct the contralateral shoulder and flex the contralateral elbow to approximately 90° while holding a 1.5 or 2 lb. hand weight. A participant will hold a 1.5 lb. hand weight if his/her body weight is less than 175 lbs., and hold a 2 lb. hand weight if his/her body weight is more than 175 lbs. First, the EMG activity of the LM was recorded during a contralateral arm lift (Figure 1a), which has been shown to best elicit LM muscle activation. A verbal instruction will be given before the participant performed the contralateral arm lift: "Breathe normally. Without moving your pelvis or spine, raise your arm above the table". Each participant will be given one practice trial before EMG recording begins, and then perform a 5-second contralateral arm lift five times. If a participant demonstrate difficulty in holding for 5 seconds, the participant will be allowed to hold for a shorter period of time, but a minimum of 3 seconds.

   Next, two trials of maximal voluntary isometric contraction (MVIC) of the LM muscles will be obtained by asking the participant to perform a contralateral arm lift while the investigator applies a steady downward force on the elbow opposite the side of the tested LM muscles (Figure 1b). Two 5-second MVIC trials will be recorded with a minimum of a 1-min rest between the two trials.
2. Pressure-pain Threshold (PPT) Testing

   For PPT testing, participants will be instructed to stop the test as soon as the "pressure" becomes "uncomfortable or painful" and will be instructed not to allow the "uncomfortable or painful sensation" to continue. A standardized instruction will be given to each participant prior to PPT testing:

   "This is a patient safety unit. (The investigator will show the participant the unit). Please hold it with the hand opposite of the testing side. When the testing begins, we will push the rounded tip of this instrument (point to the pressure algometer) into this muscle (point to the testing point) and you will feel a "pressure-like" sensation. As soon as this pressure-like sensation becomes painful or uncomfortable to you, push the green button of the patient safety unit immediately. By pushing the green button, you can stop the testing. Do not let this painful or uncomfortable sensation continue." Four trials will be performed on each of two tender points.
3. Interventions

   Three investigators are experienced physical therapists in treating patients with LBP. All are certificated manual therapists and fellows with the America Academy of Orthopedic Manual Physical Therapy. In addition, one investigator has practiced dry-needling for the past 12 years and the other two have practiced dry-needling for the past 5 years. Before data collections, the two dry-needling intervention techniques will be standardized so that all three investigators will be able to administer either one of the two dry-needling techniques when they are needed. In addition, the research assistants who will collect the outcome measures (EMG activity and PPT) will be blinded to the type of the dry-needling techniques.

   Once baseline outcome measures are collected, each participant will be randomly assigned into one of the dry-needling intervention techniques, with and without needle manipulation. The insertion of the needles will be the same for both techniques. A sterile, disposable 0.30 mm x 50 mm or 0.30 x 60 mm solid filament needle (Seirom Corp., Shizuoka, Japan) will be inserted into the bilateral LM muscles approximately 1.5 cm lateral to the L5 or S2 spinous process level. The needling sites are corresponding to the EMG and PPT testing points. The needles used in the study will be exactly the same needles used for acupuncture. After piercing the skin, the needle will be directed toward the spinous process in a slight inferior-medial angle (approximately 20 °). This angle was chosen because the needle will be stopped by the bony laminia part of vertebra to ensure a safe intervention and to standardize the depth of the needle insertion.

   For the needle manipulation technique, the needle will be pulled in and out (sparrow pecking) and redirected in small angles (coning) for 5-10 seconds. For the non-needling manipulation technique, the four needles will stay (in situ) for 10 minutes after the insertion of the needle. The investigator who administers the dry needling interventions will wear gloves during the intervention and will dispose of the used needles in a sharp container. Because needles will be used in the study, universal precautions will be followed throughout the data collection.
4. Reassessment

Immediately after the dry-needling intervention, the two outcome measures (EMG activity and PPTs) will be collected again. Each participant will also be asked about any presence of common adverse symptoms, including increased pain, nausea, dizziness and fatigue. If bleeding occurs, the participant will be informed of the occurrence. All participants will also be asked to avoid strenuous trunk activity or exercises for the following week. All participants will be scheduled to return in approximately 1 week for the final reassessment, including EMG activity and PPT testing. After return, all participants will be re-questioning about whether they experience any adverse symptoms after dry-needling.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking adults and are 18 years of age or older.
* For asymptomatic healthy adults: no existing low back pain (LBP) and no LBP in the past 6 months.
* For individuals with LBP: existing LBP near the L5-S1 level with an average pain intensity score ≥ 2/10 in the past 24 hours (numeric pain rating scale of 0-10, 0 being no pain, 10 being unbearable pain)

Exclusion Criteria (for both the asymptomatic healthy and patients with low back pain groups) :

* Bleeding disorders (e.g. hemophilia)
* Use of anti-coagulants (e.g. Coumadin)
* Previous low back surgery, systemic joint disease (e.g. rheumatoid arthritis)
* Cancer of the lower quadrant,
* Neurological disorders
* Allergic reaction to adhesive tape
* Inability to obtain testing positions (prone lying)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-09-22 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of Muscle activity | Before intervention, immediately after intervention and one week after intervention
  An electroencephalographic (EMG) system with 4 wireless surface electrodes will be used to obtain muscle activities of the right and left lumbar multifidus muscles at the L5 and S2 levels.
Change of Pressure pain threshold | Before intervention, immediately after intervention and one week after intervention
  A hand-held computerized pressure algometer will be used to determine the pressure pain threshold on the same 4 sites of EMG recording.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Wang-Price, Principal Investigator — Texas Woman's University
Locations (1):
- Texas Woman's University, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang-Price S, Zafereo J, Couch Z, Brizzolara K, Heins T, Smith L. Short-term effects of two deep dry needling techniques on pressure pain thresholds and electromyographic amplitude of the lumbosacral multifidus in patients with low back pain - a randomized clinical trial. J Man Manip Ther. 2020 Dec;28(5):254-265. doi: 10.1080/10669817.2020.1714165. Epub 2020 Jan 17. PMID 31960773